CLINICAL TRIAL: NCT03145688
Title: Promoting Habit Formation in Family Physical Activity
Brief Title: Family Habit Physical Activity Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); University of British Columbia (Other); Dalhousie University (Other); University of Alberta (Other); King's College London (Other)
Responsible Party: Principal Investigator, Ryan Rhodes, Professor, Principal Investigator, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 35941 51350
Record Dates: First submitted 2017-01-27; First posted 2017-05-09 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Physical Activity
Keywords: Behavioural; Family physical activity habit
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The control group package will consist of the Canadian 24 Hour Movement Guidelines recommending 60 minutes of moderate to vigorous physical activity per day for children. The guide also contains arguments & information about the benefits of physical activity.
- Family physical activity Planning (Experimental): Behavoural: Family Physical Activity Planning. The physical activity planning intervention condition will receive the same guidelines as the standard education control group but will also be provided with family physical activity planning material. This material will include workbook on how to plan for family physical activity; brainstorming exercises for parents & children where they list physical activities that they have found fun in the past, as well as some new activities they would like to try & skill training content to help with goal setting & tracking of physical activity.
  Interventions: Behavioral: Family Physical Activity Planning
- Family Physical Activity Habit Formation (Experimental): Behavioural: Family Physical Activity Habit formation. The Habit formation intervention condition will receive the same content as the education control condition and the physical activity planning condition but with additional material on creating physical activity support habits. The material includes a brief discussion of what habits are with some very straightforward examples such as preparing for sleep routines or initiating to drive a car to work. A key component of the habit section will be based on planning for context-dependent repetition, with pointers on how to maintain repetition as habit forms.
  Interventions: Behavioral: Family Physical Activity Habit Formation

INTERVENTIONS:
Behavioral: Family Physical Activity Planning — Families will receive the same guidelines as the standard education control group but will also be provided with family physical activity planning material. This material will include a skill training content workbook on how to plan for family physical activity. The material includes a brainstorming exercise for parents where they list physical activities they think their children have found fun in the past, as well as activities that they would find enjoyable to do as a family. We will provide this material as prompts/suggestions. Families will be instructed to plan for "when," "where," "how," and "what" physical activity will be performed & then track their physical activity. These aspects will be re-introduced and discussed at week 6 and week 12 in booster sessions
  Arms: Family physical activity Planning
Behavioral: Family Physical Activity Habit Formation — Families will receive the same content as the education control condition and the physical activity planning condition but with additional material on creating physical activity support habits. A key component of the habit section will be based on planning for context-dependent repetition, with pointers on how to maintain repetition as habit forms. The importance of creating cues for parental support of child physical activity is then outlined. Cues will also be considered factors that a) can precede the support activity but b) not be present very often when the activity is not to be performed. We will suggest that cues that have repeated exposure during times when family physical activity is not present Parents will then be asked to brainstorm and create a plan of consistency and cues with the workbooks provided. These aspects will be re-introduced and discussed at week 6 and week 12 in booster sessions.
  Arms: Family Physical Activity Habit Formation

SUMMARY:
The purpose of this study is to examine physical activity habit formation in parents and if this can increase moderate to vigorous physical activity behavior in their children over six months. The Primary Research Question is:

Does the habit formation condition result in increased moderate-vigorous intensity physical activity of the child compared to the control (education) and education + planning conditions at six months? Hypothesis: Child physical activity will be higher for the habit formation condition in comparison to the more standard physical activity education and planning conditions at six months.

DETAILED DESCRIPTION:
Secondary Research Questions

1. Does the habit formation condition improve child health-related quality of life, and health-related fitness outcomes compared to the control and planning conditions at six months? Hypothesis: Child health-related fitness and quality of life will be higher for the habit formation condition in comparison to the control and planning conditions.
2. Can group differences among behavioural, and health-related fitness outcomes be explained through a mediation model? Hypothesis: The covariance of the assigned conditions (habit formation, planning + education, education control) on child physical activity will be explained by parental support habit, and through the use of consistency and cues regulation strategies (i.e., manipulation check). In turn, the covariance between support habit and health-related outcomes will be explained by physical activity among conditions. The habit formation condition will not affect parental support intentions or underlying outcome expectations (benefits of physical activity) for support of child physical activity because its effect on behavior is to tie initial intentions to behavioural action or to work independent of goals and intentions.
3. Is there an intergenerational, seasonal, or gender difference across primary outcomes by assigned condition? Hypothesis: Parents in the habit formation condition will show higher physical activity via some activities being performed with their children in comparison to the other conditions. No differences in gender or season are hypothesized but these are exploratory research questions because there is limited research at present [28] to make any definitive statement.

ELIGIBILITY:
Inclusion Criteria:

* parents with children between the ages of 6 and 12 years
* self-report low family physical activity
* target child is not meeting Canada's Physical Activity guidelines

Exclusion Criteria:

• participant is unsafe to participate in physical activity as determined by answers to the Physical Activity Readiness Questionnaire (PAR-Q)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2017-02-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in children's physical activity to 6 months | Baseline & 6 months
  Children's physical activity will be quantified by accelerometry. Children will wear an accelerometer for a minimum of 10 hours per day for 7 days at baseline and 6 months. Additionally this measure will assess intermediate outcomes at 6 weeks and 3 months.

SECONDARY OUTCOMES:
Change from baseline in personal physical activity to six months (child PA) | Baseline & 6 months
  The target child will complete a modified version of the Physical Activity Questionnaire for Children (PAQ-C) to assess habitual moderate to vigorous physical activity. The Godin Leisure-Time Exercise Questionnaire (LSI) will be used to measure parent-reported child physical activity. Questions assess intensity, frequency, and duration of physical activity in an average week. These measures will be assessed at baseline, 6 weeks, 3 months, and 6 months.
Change from baseline in self-reported family based physical activity to six months | Baseline & 6 months
  A modified Godin Leisure-Time Exercise Questionnaire (LSI) will be used to measure parent reported family physical activity. Questions ask about frequency and duration of structured vs unstructured physical activity performed as a family. Additionally, this measure will assess intermediate outcomes at 6 weeks and 3 months
Change from baseline in weight at 6 months | baseline and 6 months
  Weight will be measured in kilograms using a scale as per standard anthropometric procedures. Change in weight will be examined from baseline to 6 months (post-intervention). Weight measurement will also contribute to change in BMI.
Change from baseline in height at 6 months | baseline and 6 months
  Height will be measured in centimeters using a stadiometer as per standard anthropometric procedures. Change in height will be examined from baseline to 6 months (post-intervention). Height measurement will also contribute to change in BMI.
Change from baseline in waist circumference at 6 months | baseline and 6 months
  Waist circumference will be measured in centimeters using a tape measuer as per standard anthropometric procedures. Change in waist circumference will be examined from baseline to 6 months (post-intervention).
Change from baseline in BMI at 6 months | baseline and 6 months
  Change in BMI will be examined from baseline to 6 months (post intervention) using height and weight measurements in the following formula: (weight in kg)/(height in meters)^2.
Change from baseline in grip strength at 6 months (MSK fitness) | baseline and 6 months
  Grip strength of the target child will be measured using the Canadian CSEP standardized protocols. Change in grip strength from baseline to 6 months (i.e., post-intervention) will be examined
Change from baseline in sit and reach flexibility at 6 months | baseline and 6 months
  Sit and reach flexibility of the target child will be measured using the Canadian CSEP standardized protocols. Change in sit and reach flexibility from baseline to 6 months (i.e., post-intervention) will be examined
Change from baseline in plank test time at 6 months | baseline and 6 months
  Sit and reach flexibility of the target child will be measured using the Canadian CSEP standardized protocols. Change in plank test time from baseline to 6 months (i.e., post-intervention) will be examined
Change from baseline in cardiovascular fitness at 6 months | baseline and 6 months
  The Leger Shuttle Run will be used to assess cardiovascular fitness for target child. Change in cardiovascular fitness from baseline to 6 months (i.e., post-intervention) will be examined.
Change from baseline in parent support of child's physical activity at 6 weeks | baseline and 6 weeks
  The Activity Support Scale for Multiple Groups (ACTS-MG) will be used to measure parent support of child PA.
Change from baseline in parent support of child's physical activity at 3 months | baseline and 3 months
  The Activity Support Scale for Multiple Groups (ACTS-MG) will be used to measure parent support of child PA.
Change from baseline in parent support of child's physical activity at 6 months | baseline and 6 months
  The Activity Support Scale for Multiple Groups (ACTS-MG) will be used to measure parent support of child PA.
Change from baseline in parent support habits of child physical activity at 6 months (a) | baseline and 6 months
  Self report habit strength index will be used to measure parental support habit for child Physical Activity. This tool measures habit strength and automaticity at baseline, 6 weeks, 3 months and 6 months.

OTHER OUTCOMES:
TERTIARY OUTCOME - Change from baseline in personal physical activity to 6 months (parent) | Baseline and 6 months
  Tertiary Outcome Measure The Godin Leisure-Time Exercise Questionnaire (LSI) will be used to measure self - reported physical activity at baseline, 6 weeks, 3 months, 6 months. Questions assess intensity, frequency, and duration of physical activity in an average week.
TERTIARY OUTCOME - Change from baseline in health-related quality of life at 6 months | baseline & 6 months
  Tertiary Outcome Measure Quality of life will be assessed with parents using the 12 item Short Form Health Survey. Scores can range from 0-100 with a higher score indicating better health. Change in health-related quality of life from baseline to 6 months (i.e., post-intervention) will be examined with intermediate time points of 6 weeks and 3 months as well.
TERTIARY OUTCOME - Change from baseline in family functioning at 6 months | baseline and 6 months
  Tertiary Outcome Measure Family Environment Scale is used to assess family functioning at baseline, 6 weeks, 3 months, and 6 months. Total score can range from 0 (total agreement between family members) to 90 (total disagreement between family members).
TERTIARY OUTCOME - Change from baseline in motivations (MPAC constructs) at 6 weeks | baseline & 6 weeks
  Tertiary Outcome Measure Motivations for supporting child based physical activity will be measured using the constructs of the Theory of Planned Behaviour & Self Determination Theory including affective attitude, instrumental attitude, perceived behavioural control, behavioural regulation, intention, and identity. These measures are all part of the Multi Process Action Control Framework (MPAC).
TERTIARY OUTCOME - Change from baseline in motivations (MPAC constructs) at 3 months | baseline and 3 months
  Tertiary Outcome Measure Motivations for supporting child based physical activity will be measured using the constructs of the Theory of Planned Behaviour & Self Determination Theory including affective attitude, instrumental attitude, perceived behavioural control, behavioural regulation, intention, and identity. These measures are all part of the Multi Process Action Control Framework (MPAC).
TERTIARY OUTCOME - Change from baseline in motivations (MPAC constructs) at 6 months | baseline and 6 months
  Tertiary Outcome Measure Motivations for supporting child based physical activity will be measured using the constructs of the Theory of Planned Behaviour & Self Determination Theory including affective attitude, instrumental attitude, perceived behavioural control, behavioural regulation, intention, and identity. These measures are all part of the Multi Process Action Control Framework (MPAC).
Change from baseline to 6 months in cue consistency (manipulation check) | Baseline and 6 months
  Cue consistency will be assessed using a 6 item survey. Answers range from not at all true (1) to very true (7) with a higher score indicating greater cue consistency. Changes in cue consistency will be examined at 6 months with intermediate time points of 6 weeks and 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Rhodes, PhD, Principal Investigator — University of Victoria; Chris Blanshard, PhD, Study Chair — Dalhousie University; Valerie Carson, PhD, Study Chair — University of Alberta; Benjamin Gardner, PhD, Study Chair — King's College London; Darren Warburton, PhD, Study Chair — University of British Columbia; Mark Beauchamp, PhD, Study Chair — University of British Columbia
Locations (1):
- Behavioural Medicine Lab, University of Victoria, Victoria, British Columbia, Canada

REFERENCES:
- [Derived] Medd ER, Beauchamp MR, Blanchard CM, Carson V, Gardner B, Warburton DE, Rhodes RE. Family-based habit intervention to promote parent support for child physical activity in Canada: protocol for a randomised trial. BMJ Open. 2020 Apr 14;10(4):e033732. doi: 10.1136/bmjopen-2019-033732. PMID 32295773